CLINICAL TRIAL: NCT06625216
Title: Observatory of Patients with Severe Asthma and Potential Eligible Patients for Treatment with Biological Drugs
Brief Title: Severe Asthma Network Italy
Acronym: SANI
Status: Recruiting | Type: Observational
Sponsor: Società Italiana di Allergologia, Asma e Immunologia Clinica (Other)
Collaborators: Societa Italiana di Pneumologia (Other)
Responsible Party: Sponsor
Other Study IDs: ICH 1742
Record Dates: First submitted 2024-07-05; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Severe Asthma
Keywords: Severe Asthma; Network; Registry; Biologics; Adherence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and induced sputum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this registry is collecting data of severe asthma patients, recruited by specialized centers, in a real life setting, homogeneously placed on a database management system to follow them over the time.

The information recorded will provide:

1. The collection of homogeneous clinical, functional and biologic data of patients with severe asthma in a real life setting.
2. The evaluation of adherence to treatment in real life.
3. The clinical eligibility of patients treated with biologics.
4. The evaluation of patients' clinical response to each treatment.
5. The monitoring of tolerability and safety.
6. The long-term follow up of patients with severe asthma.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent and privacy disclaimer;
2. age > 12 years;
3. diagnosis of severe asthma according to the ERS/ATS criteria:

   1. During treatment with:

      * High-dose ICS + at least one addistional controller (LABA, montelukast, or theophylline) or
      * Oral corticosteroids >6 months/year
   2. at least one of the following occurs or would occur if treatment would be reduced:

      * ACT <20 or ACQ>1.5
      * At least 2 exacerbations in the last 12 months
      * At least 1 exacerbation treated in hospital or requiring mechanical ventilation in the last 12 months
      * FEV1 <80% (if FEV1/FVC below the lower limit of normal)

Exclusion Criteria have not been considered in order to have a realistic view of severe asthma in real life.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 12 years, diagnosed for severe asthma by a specialist, according to the ERS/ATS criteria, attending respiratory or allergy clinic for a scheduled visit are eligible for study enrollment. If inclusion/exclusion criteria are satisfied, a written consent to participate in the study will be obtained and an informative leaflet for the patient and his/her GPs will be delivered.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-02-17 (Actual); Primary Completion 2027-02-17 (Estimated); Study Completion 2037-02-17 (Estimated)

PRIMARY OUTCOMES:
Analyzing epidemiological and clinical characteristics of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Collection of sociodemographic data: sex, employment, ethnicity, smocking habits.
Analyzing epidemiological and clinical characteristics of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Collection of clinical data: age, age at asthma onset and/or age at asthma diagnosis (years).
Analyzing epidemiological and clinical characteristics of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Collection of clinical data: weight (kilograms) and height (meters) combined to report Body Mass Index [BMI] in kg/m^2.
Analyzing epidemiological and clinical characteristics of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Collection of clinical data: presence of allergies and/or comorbidities, previous accesses to ER and/or hospitalizations, and numbers of exacerbations.
Collecting functional data of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Assessment of lung function before and after a bronchodilator medication: Forced Vital Capacity [FVC] and Forced Expiratory Volume in 1 second [FEV1] values (liters) combined to report FEV1/FVC Ratio.
Collecting functional data of severe asthmatics from SANI registry. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Assessment of lung function before and after a bronchodilator medication: Forced Vital Capacity [FVC] and Forced Expiratory Volume in 1 second [FEV1] values (percentages) combined to report FEV1/FVC Ratio.
Assessing inflammatory markers in order to characterize asthma endotypes. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Measurement of Fractional exhaled Nitric Oxide [FeNO] (ppb).
Assessing inflammatory markers in order to characterize asthma endotypes. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Measurement of total serum IgE (kU/L).
Assessing inflammatory markers in order to characterize asthma endotypes. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Measurement of blood eosinophilia (10^9 cells/L).
Assessing inflammatory markers in order to characterize asthma endotypes. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Measurement of blood and sputum eosinophil levels (percentages).
Assessing asthma control and and PROs. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Assessment of asthma control over time according to the GINA Guidelines and standardized questionnaires: Asthma Control Test [ACT], and Asthma Control Questionnaire [ACQ].
Assessing asthma control and and PROs. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Assessment of the quality of life through Asthma Quality of Life Questionnaire [AQLQ] .
Studying the real life efficacy and safety of biologics. | through study completion (the length of the follow up for each patient is scheduled for 10 years)
  Evaluation of patients' clinical response to each biologics, reports of previous adverse reactions to the drug used and reasons for withdrawal from biologic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Marco Heffler, MD, PhD, Study Chair — Personalized Medicine, Asthma and Allergy - IRCCS Humanitas Research Hospital, Rozzano, Italy
Locations (1):
- Personalized Medicine, Asthma and Allergy - IRCCS Humanitas Research Hospital, Rozzano, Italy, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wenzel S. Severe asthma: from characteristics to phenotypes to endotypes. Clin Exp Allergy. 2012 May;42(5):650-8. doi: 10.1111/j.1365-2222.2011.03929.x. Epub 2012 Jan 18. PMID 22251060
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] De Ferrari L, Chiappori A, Bagnasco D, Riccio AM, Passalacqua G, Canonica GW. Molecular phenotyping and biomarker development: are we on our way towards targeted therapy for severe asthma? Expert Rev Respir Med. 2016;10(1):29-38. doi: 10.1586/17476348.2016.1111763. Epub 2015 Nov 13. PMID 26566089
- [Background] Latorre M, Baldini C, Seccia V, Pepe P, Novelli F, Celi A, Bacci E, Cianchetti S, Dente FL, Bombardieri S, Paggiaro P. Asthma Control and Airway Inflammation in Patients with Eosinophilic Granulomatosis with Polyangiitis. J Allergy Clin Immunol Pract. 2016 May-Jun;4(3):512-9. doi: 10.1016/j.jaip.2015.12.014. Epub 2016 Feb 13. PMID 26883543
- [Background] Chung KF. Targeting the interleukin pathway in the treatment of asthma. Lancet. 2015 Sep 12;386(9998):1086-96. doi: 10.1016/S0140-6736(15)00157-9. PMID 26383000
- [Background] Pelaia G, Vatrella A, Maselli R. The potential of biologics for the treatment of asthma. Nat Rev Drug Discov. 2012 Dec;11(12):958-72. doi: 10.1038/nrd3792. PMID 23197041
- [Background] Bagnasco D, Ferrando M, Bernardi S, Passalacqua G, Canonica GW. The path to personalized medicine in asthma. Expert Rev Respir Med. 2016 Sep;10(9):957-65. doi: 10.1080/17476348.2016.1205490. Epub 2016 Jul 11. PMID 27399975
- [Background] Chipps BE, Zeiger RS, Dorenbaum A, Borish L, Wenzel SE, Miller DP, Hayden ML, Bleecker ER, Simons FE, Szefler SJ, Weiss ST, Haselkorn T; TENOR Study Group. Assessment of asthma control and asthma exacerbations in the epidemiology and natural history of asthma: outcomes and treatment regimens (TENOR) observational cohort. Curr Respir Care Rep. 2012 Dec;1(4):259-269. doi: 10.1007/s13665-012-0025-x. Epub 2012 Sep 20. PMID 23136642
- [Background] Chipps BE, Zeiger RS, Borish L, Wenzel SE, Yegin A, Hayden ML, Miller DP, Bleecker ER, Simons FE, Szefler SJ, Weiss ST, Haselkorn T; TENOR Study Group. Key findings and clinical implications from The Epidemiology and Natural History of Asthma: Outcomes and Treatment Regimens (TENOR) study. J Allergy Clin Immunol. 2012 Aug;130(2):332-42.e10. doi: 10.1016/j.jaci.2012.04.014. Epub 2012 Jun 12. PMID 22694932
- [Background] Schleich F, Brusselle G, Louis R, Vandenplas O, Michils A, Pilette C, Peche R, Manise M, Joos G. Heterogeneity of phenotypes in severe asthmatics. The Belgian Severe Asthma Registry (BSAR). Respir Med. 2014 Dec;108(12):1723-32. doi: 10.1016/j.rmed.2014.10.007. Epub 2014 Oct 27. PMID 25456708
- [Background] Ferry JJ, Horvath AM, Bekersky I, Heath EC, Ryan CF, Colburn WA. Relative and absolute bioavailability of prednisone and prednisolone after separate oral and intravenous doses. J Clin Pharmacol. 1988 Jan;28(1):81-7. doi: 10.1002/j.1552-4604.1988.tb03105.x. PMID 3350994
- [Background] Normansell R, Walker S, Milan SJ, Walters EH, Nair P. Omalizumab for asthma in adults and children. Cochrane Database Syst Rev. 2014 Jan 13;2014(1):CD003559. doi: 10.1002/14651858.CD003559.pub4. PMID 24414989
- [Background] Novelli F, Latorre M, Vergura L, Caiaffa MF, Camiciottoli G, Guarnieri G, Matucci A, Macchia L, Vianello A, Vultaggio A, Celi A, Cazzola M, Paggiaro P; Xolair Italian Study Group. Asthma control in severe asthmatics under treatment with omalizumab: a cross-sectional observational study in Italy. Pulm Pharmacol Ther. 2015 Apr;31:123-9. doi: 10.1016/j.pupt.2014.09.007. Epub 2014 Sep 30. PMID 25281265
- [Background] Caminati M, Senna G, Guerriero M, Dama AR, Chieco-Bianchi F, Stefanizzi G, Montagni M, Ridolo E. Omalizumab for severe allergic asthma in clinical trials and real-life studies: what we know and what we should address. Pulm Pharmacol Ther. 2015 Apr;31:28-35. doi: 10.1016/j.pupt.2015.01.006. Epub 2015 Jan 30. PMID 25640019
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Braunstahl GJ, Chen CW, Maykut R, Georgiou P, Peachey G, Bruce J. The eXpeRience registry: the 'real-world' effectiveness of omalizumab in allergic asthma. Respir Med. 2013 Aug;107(8):1141-51. doi: 10.1016/j.rmed.2013.04.017. Epub 2013 May 28. PMID 23721684
- [Background] Rodrigo GJ, Neffen H, Castro-Rodriguez JA. Efficacy and safety of subcutaneous omalizumab vs placebo as add-on therapy to corticosteroids for children and adults with asthma: a systematic review. Chest. 2011 Jan;139(1):28-35. doi: 10.1378/chest.10-1194. Epub 2010 Aug 5. PMID 20688929
- [Background] Omalizumab Treatment for Adults and Children with Allergic Asthma: A Review of the Clinical Effectiveness, Cost-Effectiveness, and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2015 Mar 9. Available from http://www.ncbi.nlm.nih.gov/books/NBK280029/ PMID 25834884
- [Derived] Ridolo E, Ottoni M, Nicoletta F, Locatelli F, Martinelli L, Maule M, Cheema NA, Blasi F, Paggiaro P, Heffler E, Brussino L, Canonica GW, Senna G, Caminati M; SANI network. Role of body anthropometry in severe asthmatic patients: Evidences from the Severe Asthma Network in Italy (SANI) registry. World Allergy Organ J. 2025 May 5;18(5):101056. doi: 10.1016/j.waojou.2025.101056. eCollection 2025 May. PMID 40458738
- [Derived] Canonica GW, Blasi F, Paggiaro P, Heffler E, Braido F, Brussino L, Scioscia G, Cardini C, Oriecuia C, Sala I, Bagnardi V; SANI (Severe Asthma Network in Italy) study group. Biologics as well as inhaled anti-asthmatic therapy achieve clinical remission: Evidence from the Severe Asthma Network in Italy (SANI). World Allergy Organ J. 2024 Dec 27;18(1):101016. doi: 10.1016/j.waojou.2024.101016. eCollection 2025 Jan. PMID 39829953
- See also: Global Initiative for Asthma (GINA). Global Strategy for Asthma Management and Prevention, Revised 2014. Global Initiative for Asthma 2014 — http://www.ginasthma.org